CLINICAL TRIAL: NCT01194856
Title: A Randomized Study to Evaluate the Effect of Switching From Efavirenz to Atazanavir/ Ritonavir on Lipoatrophy and Mitochondrial Dysfunction in HIV-infected Subjects With Good Virologic Suppression
Brief Title: Switching From Efavirenz to Atazanavir/ Ritonavir in HIV-infected Subjects With Good Virologic Suppression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Closed due to low enrollment
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Case Western Reserve University (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Marisa Tungsiripat, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-418; 5K23AI070078 (NIH); BMS100MT (Other Grant/Funding Number: Bristol Myers Squibb)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: HIV Infection; Mitochondrial Dysfunction
Keywords: HIV; Lipoatrophy; mitochondrial dysfunction
MeSH Terms: conditions — HIV Infections; Mitochondrial Diseases; Lipodystrophy | interventions — atazanavir, ritonavir drug combination; Atazanavir Sulfate; Ritonavir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efavirenz 600 mg (Active Comparator): Serving as the Control Arm - patients will maintain EFV-containing antiretroviral regimen
  Interventions: Drug: Efavirenz
- Arm B - Atazanavir/Ritonavir (Experimental): Atazanavir 300 mg orally with Ritonavir 100 mg orally once daily for 96 wks
  Interventions: Drug: Atazanavir/ritonavir

INTERVENTIONS:
Drug: Atazanavir/ritonavir — 300 mg orally once daily with Ritonavir 100mg orally once daily for 96 weeks
  Other Names: Reyataz®: 100 mg, 150 mg, 200 mg, 300 mg; Norvir®: 100 mg
  Arms: Arm B - Atazanavir/Ritonavir
Drug: Efavirenz — Maintain dosage - 600 mg orally QHS for 96 weeks
  Other Names: Sustiva®: 50 mg, 200 mg
  Arms: Efavirenz 600 mg

SUMMARY:
The purposes of this study are to evaluate if switching an antiretroviral medication from efavirenz (EFV) to atazanavir/ ritonavir (ARV/r) will, in a 96-week period, change:

1. the amount of fat in HIV patients with lipoatrophy,
2. metabolic lab values such as your lipid (fat) profile, glucose (blood sugar), and insulin (a hormone that regulates glucose) in HIV patients with lipoatrophy.

DETAILED DESCRIPTION:
Our study will evaluate the effects on peripheral fat of switching from EFV to ATV/r over 96 weeks in HIV+ patients with clinical lipoatrophy. From a virologic standpoint, EFV and ATV/r are medications which are recommended equally as preferred components of antiretroviral regimens in the December 2009 version of the Guidelines for the Use of Antiretroviral Agents in HIV-1 Infected Adults and Adolescents.[20] The study subjects should be receiving a stable EFV-containing antiretroviral (ART) regimen for at least 48 weeks prior to study entry. Blood will be saved for further investigations if needed. Safety parameters will be regularly assessed throughout the study. In addition, a subcutaneous fat biopsy will be obtained to measure fat mtDNA, mtRNA, and fat apoptosis. These measurements would provide significant insight into the clinical changes which have been recently described.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection
2. Age > or = 18 years old.
3. Signed informed consent.
4. Clinical lipoatrophy of at least moderate severity and in at least two different areas of the following: face, arms, legs, or buttocks (as self reported by the patient and confirmed by the physician).
5. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.
6. All subjects must not participate in a conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female subject/ male partner must use condoms (male or female) in addition to one of the following forms of contraception while on study: either a spermicidal agent, diaphragm, cervical cap, IUD, or hormonal-based contraception.

   Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
7. Receiving EFV-containing antiretroviral regimen for at least the last 48 weeks prior to study entry. Backbone NRTI regimens can include tenofovir, abacavir, emtricitabine, and/ or lamivudine. Backbone NRTI regimens cannot include zidovudine, stavudine, or didanosine. Breaks in therapy for a maximum of 5 consecutive days will be allowed during these 48 weeks, including the period immediately preceding study entry.
8. Patient willing and able to stop aspirin/ NSAIDS for 7 days before study entry and the scheduled skin biopsy procedures.
9. HIV-1 RNA < 400 copies/mL for at least 90 days prior to study entry.
10. Laboratory values obtained within 60 days prior to study entry:

    1. Absolute neutrophil count (ANC) ≥ 500 / mm3
    2. Hemoglobin ≥ 9.0 g/dL
    3. Platelet count ≥ 75,000/ mm3
    4. Creatinine clearance > 50 mL / min
    5. PT/PTT < 1.2 ULN

Exclusion Criteria:

1. Receipt of AZT, d4T, ddI, or ddC at study entry or within 24 weeks of entry
2. Life expectancy < 12 months
3. Women who are pregnant or breastfeeding
4. WOCBP unwilling to use contraception WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
5. Women with a positive pregnancy test.
6. Sexually active fertile men not using effective birth control if their partners are WOCBP.
7. Other Exclusion Criteria

   1. Prisoners or subjects who are involuntarily incarcerated.
   2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
8. Clinically important illness within 14 days prior to study entry
9. Inability to communicate effectively with the study personnel.
10. Bleeding diathesis
11. Supplementation with recombinant growth hormone, growth hormone releasing factor, anabolic steroids, estrogen or testosterone, unless it is for replacement purposes.
12. Have no plans to alter any vitamin supplementation that subjects are receiving at study entry. This includes all vitamin supplementation, coenzyme Q, N acetyl cysteine, L-acetyl carnitine, and uridine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Tungsiripat, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in DEXA-measured Limb Fat Between the EFV and ATV/r Arms
Description: To examine the effect of switching from EFV- to ATV/r on limb fat in HIV-1 infected patients with established lipoatrophy, the primary objective of this trial will be to compare changes over 48 weeks in DEXA-measured limb fat between the EFV arm and ATV/r.
Time Frame: 48 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare Changes for DEXA-measured Limb Fat Between EFV and ATV/r Arms
Description: To examine the effect of switching from EFV- to ATV/r on limb fat in HIV-1 infected patients with established lipoatrophy, a secondary objective of this trial will be to compare changes over 96 weeks in DEXA-measured limb fat between the EFV arm and ARV/r.
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Compare Changes in CD4, HIV-1 RNA Levels and Adverse Events in Two Arms
Description: To examine the effect of switching from EFV to ATV/r on safety in HIV-1 infected patients, a secondary objective of this trial will be to compare changes over 96 weeks in CD4 cell count, HIV-1 RNA levels, and adverse events between the EFV arm and the ATV/r arm
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Compare Changes in Fat mtDNA, mtRNA and Fat Apoptosis Between the Two Arms
Description: To examine the effect of switching from EFV to ATV/r on fat mtDNA, mtRNA, and fat apoptosis in HIV-1 infected patients, a secondary objective of this trial will be to compare changes over 96 weeks in fat mtDNA, mt RNA levels and fat apoptosis between the EFV arm and ARV/r arm.
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Comparing Fasting Lipid Levels Between the Two Arms
Description: To examine the effect of switching from EFV to ATV/r on lipids in HIV-1 infected patients, a secondary objective of this trial will be to compare changes over 96 weeks in fasting lipid levels between the EFV arm and ATV/r arm.
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Comparing Glucose Metabolism (Fasting Insulin, QUIKI and HOMA-IR) Between the Two Arms
Description: To examine the effect of switching from EFV to ATV/r on glucose metabolism in HIV-1 infected patients, a secondary objective of this trial will be to compare changes over 96 weeks in fasting insulin, QUIKI and HOMA-IR between the EFV arm and the ATV/r arm
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Compare Changes in Levels of Hs-CRP Between the Two Arms
Description: To examine the effect of switching from EFV to ATV/r on highly sensitive C-reactive protein (hs-CRP) in HIV-1 infected patients, a secondary objective of this trial will be to compare changes over 96 weeks in hs (highly sensitive) - CRP levels between the EFV arm and the ATV/r arm.
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlate the Changes in DEXA-measured Fat Limb With Fat mtDNA, mtRNA and Fat Apoptosis
Description: A secondary objective of this trial will be to correlate the changes in DEXA-measured limb fat with those of fat mtDNA, mtRNA levels and fat apoptosis
Time Frame: 96 weeks
Population: Data not collected for analysis due to low enrollment and participant discontinuation.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: We utilized the same definitions of adverse event and serious adverse event as clinicaltrials.gov.
  All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for Arm B due to no participants being randomized to that arm of the study.
Arm/Group | Efavirenz 600 mg | Arm B - Atazanavir/Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Data not collected for analysis due to low enrollment and participant discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes